CLINICAL TRIAL: NCT01755455
Title: Iron Supplementation for the Hypoferremic Anemia of Cystic Fibrosis
Brief Title: Does a Daily Iron Tablet Improve Anemia in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Alex H. Gifford, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D11176; CPHS#22884 (Other Grant/Funding Number: The Flatley Foundation)
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Anemia, Iron-Deficiency
Keywords: Cystic fibrosis; Iron; Hepcidin; Anemia; Erythropoiesis
MeSH Terms: conditions — Cystic Fibrosis; Anemia, Iron-Deficiency; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous sulfate 325mg (Active Comparator): Ferrous sulfate 325mg tablet taken by mouth daily for 6 weeks
  Interventions: Drug: Ferrous sulfate 325mg
- Placebo (Placebo Comparator): Identical-appearing tablet taken by mouth daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferrous sulfate 325mg — Ferrous sulfate 325mg tablet taken by mouth daily for 6 weeks
  Arms: Ferrous sulfate 325mg
Drug: Placebo — Matching placebo capsule
  Arms: Placebo

SUMMARY:
This study questions whether low-dose ferrous sulfate taken by mouth daily for 6 weeks increases hemoglobin concentration in adult subjects with cystic fibrosis and hypoferremic anemia.

ELIGIBILITY:
Inclusion Criteria:

* History of Pseudomonas aeruginosa colonization of the lung
* Transferrin saturation (TSAT) less than or equal to 21%
* Hemoglobin concentration <15.5 gm/dl (men)
* Hemoglobin concentration <13.6 gm/dl (women)

Exclusion Criteria:

* Use of iron-containing vitamin or supplement
* Pregnancy
* Lactation
* Cirrhosis
* History of chronic visible (gross) hemoptysis
* Hereditary hemochromatosis
* History of transfusion-related iron overload
* Use of iron chelator(s)
* Withdrawal of informed consent
* Contraindication to phlebotomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Gifford, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Maine Medical Center, Portland, Maine
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Result] Gifford AH, Alexandru DM, Li Z, Dorman DB, Moulton LA, Price KE, Hampton TH, Sogin ML, Zuckerman JB, Parker HW, Stanton BA, O'Toole GA. Iron supplementation does not worsen respiratory health or alter the sputum microbiome in cystic fibrosis. J Cyst Fibros. 2014 May;13(3):311-8. doi: 10.1016/j.jcf.2013.11.004. Epub 2013 Dec 13. PMID 24332997
- See also: Pubmed Entry — http://www.ncbi.nlm.nih.gov/pubmed/24332997

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Ferrous Sulfate: Placebo administered daily for 6 week followed by 4-week washout, then Ferrous Sulfate 325 mg administered daily for 6 weeks.
- Ferrous Sulfate, Then Placebo: Ferrous Sulfate 325 mg administered daily for 6 weeks followed by 4-week washout, then Placebo administered daily for 6 weeks.
Period: First Intervention (6 Weeks)
Arm/Group | Placebo, Then Ferrous Sulfate | Ferrous Sulfate, Then Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Placebo, Then Ferrous Sulfate | Ferrous Sulfate, Then Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Placebo, Then Ferrous Sulfate | Ferrous Sulfate, Then Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes those who started the study with First Intervention and those who started the study with Second Intervention
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (13.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin Concentration (gm/dl)
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: gm/dl
Groups:
- Placebo: Outcome measure in all participants who received placebo.
- Ferrous Sulfate: Outcome measure in all participants who received ferrous sulfate.
Arm/Group | Placebo | Ferrous Sulfate
Number analyzed (Participants) | 22 | 22
gm/dl | 0.12 (0.13) | 0.09 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Ferrous Sulfate; Fixed-effect models accounted for repeated measurements within subjects and treatment sequence. The estimated effect signifies the absolute change from baseline at 6 weeks in the specified outcome measure and (standard error); Test type: Superiority or Other; p = 0.81, Fixed-effect model

2. Secondary Outcome: Change From Baseline in Serum Iron (mcg/dl)
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: mcg/dl
Arm/Group | Placebo | Ferrous Sulfate
Number analyzed (Participants) | 22 | 22
mcg/dl | 13.7 (5.9) | -4.2 (5.7)
Statistical Analysis 1: Comparison: Placebo vs Ferrous Sulfate; Test type: Superiority or Other; p < 0.05, Fixed-effect model

3. Secondary Outcome: Change From Baseline in Transferrin Saturation (%)
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: % saturation
Arm/Group | Placebo | Ferrous Sulfate
Number analyzed (Participants) | 22 | 22
% saturation | 4.7 (1.5) | -1.8 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Ferrous Sulfate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Fixed-effect model

4. Secondary Outcome: Change From Baseline in Sputum Iron (ng/mg)
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: ng/mg
Arm/Group | Placebo | Ferrous Sulfate
Number analyzed (Participants) | 22 | 22
ng/mg | 0.13 (0.17) | 0.42 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Ferrous Sulfate; Test type: Superiority or Other; p = 0.16, Fixed-effect model

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Placebo: Events observed among all participants while they were receiving placebo.
- Ferrous Sulfate: Events observed among all participants while they were receiving ferrous sulfate.
Arm/Group | Placebo | Ferrous Sulfate
Serious Adverse Events (participants affected / at risk) | 4/22 | 3/22
Other Adverse Events (participants affected / at risk) | 13/22 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Ferrous Sulfate (N=22)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Ferrous Sulfate (N=22)
Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 11 (14)

LIMITATIONS AND CAVEATS:
The power to detect changes in Akron PES was 42%; 160 subjects would be needed to ensure that exacerbation risk was lower for ferrous sulfate with 80% power and p <0.05.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No